CLINICAL TRIAL: NCT00701831
Title: Assessment of Forced Titration to Reach the Effective Dose for Good Glycemic Control in Lantus Treated Type 2 Patients
Brief Title: Assessment of Insulin Glargine in Type 2 Patients for Good Glycemic Control
Acronym: LANTIT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Trial Transparency Team, sanofi-aventis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LANTU_L_03502
Record Dates: First submitted 2008-06-18; First posted 2008-06-19 (Estimated); Last update posted 2010-11-04 (Estimated); Status verified 2010-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

ARMS (1):
- 1 (Experimental): Insulin glargine
  Interventions: Drug: Insulin glargine

INTERVENTIONS:
Drug: Insulin glargine — The dose is titrated according to patient needs

SUMMARY:
Primary objective:

* To observe the efficacy of the forced titration to reach good glycemic control in Lantus treated patients

Secondary objectives:

* To assess the forced titration on physician and patient satisfaction
* To evaluate the impact of training tools by means of patient profile

ELIGIBILITY:
Inclusion Criteria:

* T2 insulin naïve patients
* Patients whom their physician is considering initiation of Lantus treatment
* Poor glycemic control 7,5 %10 %
* T2 treatment with OADs more than 3 months
* BMI<40 kg/m2

Exclusion Criteria:

* Impaired renal function (Cr>2mg/dl or current renal dialysis)
* Acute or chronic metabolic acidosis
* Active liver disease or serum ALT or AST >2,5 than normal
* History of hypoglycemia unawareness
* Diabetic retinopathy with surgery in the previous 3 months or planned within 3 months after study entry
* Pregnancy, breast feeding

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2008-05; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
HbA1c, FBG | after treatment end (6 months)
Final dose | after treatment end (6 months)
Number of dose adjustment | after treatment end (6 months)
Time to dose titration | after treatment end (6 months)

SECONDARY OUTCOMES:
Hypoglycemia | after treatment end (6 months)
Noctural hypoglycemia | after treatment end (6 months)
DTSQ | after treatment end (6 months)
Physician Satisfaction Questionnaire | after treatment end (6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Cetin, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Istanbul, Turkey (Türkiye)